CLINICAL TRIAL: NCT01214850
Title: A Phase 3 Observer Blind Randomized, Multi-center, Controlled Study to Evaluate the Effect of Novartis Vaccine's Meningococcal B Recombinant and MenACWY Conjugate Vaccines on Pharyngeal Carriage of N. Meningitidis in Young Adults
Brief Title: Novartis Vaccine and Diagnostics Carriage Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V72_29
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: N. Meningitidis Carriage
Keywords: Meningococcal vaccines; Meningococcal B; Meningococcal ACWY serogroups
MeSH Terms: interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- rMenB+OMV (Experimental): Subjects (18-24 years) received two injections of rMenB+OMV NZ vaccine, one month apart
  Interventions: Biological: Meningococcal B Recombinant + Outer Membrane Vesicle vaccine (rMenB+OMV NZ)
- MenACWY (Experimental): Subjects (18-24 years) received one injection of MenACWY-CRM vaccine followed by one injection of placebo, one month apart
  Interventions: Biological: MenACWY-CRM conjugate vaccine
- Control (Active Comparator): Subjects (18-24 years) received two injections of a control vaccine (Japanese Encephalitis), one month apart
  Interventions: Biological: Japanese Encephalitis vaccine

INTERVENTIONS:
Biological: Meningococcal B Recombinant + Outer Membrane Vesicle vaccine (rMenB+OMV NZ)
  Arms: rMenB+OMV
Biological: MenACWY-CRM conjugate vaccine
  Arms: MenACWY
Biological: Japanese Encephalitis vaccine
  Other Names: IXIARO
  Arms: Control

SUMMARY:
The purpose of this trial was to evaluate the effect of Novartis Vaccine's Meningococcal vaccines on carriage of Neisseria meningitidis in a young adult population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, 18-24 years of age who provided written informed consent at the time of enrollment;
* Subjects who were available for all the visits scheduled in the study;
* Subjects who were in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

* History of any serogroup B meningococcal vaccine administration;
* Current or previous, confirmed or suspected disease caused by N. meningitidis;
* Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment;
* Significant acute or chronic infection within the previous 7 days or fever (defined as oral temperature ≥38ºC) within the previous day;
* Antibiotics within 3 days (72 hours) prior to enrollment;
* Pregnancy or nursing (breastfeeding) mothers;
* Females of childbearing age who had not used or did not plan to use acceptable birth control measures, for the 12 months duration of the study. Oral, injected or implanted hormonal contraceptive, diaphragm, condom, intrauterine device or sexual abstinence were considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods for at least 30 days prior to study entry;
* Any serious chronic or progressive disease (e.g., neoplasm, diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition);
* Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, including use of corticosteroids in immunosuppressive doses or chronic use of inhaled high-potency corticosteroids within the previous 60 days. [Use of topical corticosteroids administered during the study in limited areas (i.e., eczema on knees or face or elbows) of the body were allowed]; use of immunostimulants;
* Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
* Participation in another clinical trial within the last 90 days or planned for during study;
* Family members and household members of research staff;
* Any condition which in the opinion of the investigator and/or the Regional MD may interfere with the evaluation of the study objectives.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2968 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (10):
- United Kingdom (10):
  - Clinical Research Center, University of Surrey, Surrey, England
  - Bristol Children's Vaccine Center, University of Bristol,, Bristol, England
  - Royal Liverpool and Broad Green University Hospital Trust, Liverpool, England
  - St Georges Vaccine Institute, St Georges, University of London, London, England
  - Manchester Welcome Trust Clinical Research Facility, University of Manchester, Manchester, England
  - The James Cook University Hospital, Middlesbrough, England
  - Cripps Health Centre, University Park, Nottingham, England
  - University of Oxford, Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, England
  - Clinical Research Facility, Royal Hallamshire Hospital, Sheffield, England
  - Wellcome Trust Clinical Research Facility, University of Southampton, Southampton, England

REFERENCES:
- [Derived] Lemee L, Hong E, Etienne M, Deghmane AE, Delbos V, Terrade A, Berthelot G, Caron F, Taha MK. Genetic diversity and levels of expression of factor H binding protein among carriage isolates of Neisseria meningitidis. PLoS One. 2014 Sep 23;9(9):e107240. doi: 10.1371/journal.pone.0107240. eCollection 2014. PMID 25247300
- [Derived] Read RC, Baxter D, Chadwick DR, Faust SN, Finn A, Gordon SB, Heath PT, Lewis DJ, Pollard AJ, Turner DP, Bazaz R, Ganguli A, Havelock T, Neal KR, Okike IO, Morales-Aza B, Patel K, Snape MD, Williams J, Gilchrist S, Gray SJ, Maiden MC, Toneatto D, Wang H, McCarthy M, Dull PM, Borrow R. Effect of a quadrivalent meningococcal ACWY glycoconjugate or a serogroup B meningococcal vaccine on meningococcal carriage: an observer-blind, phase 3 randomised clinical trial. Lancet. 2014 Dec 13;384(9960):2123-31. doi: 10.1016/S0140-6736(14)60842-4. Epub 2014 Aug 18. PMID 25145775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 10 sites in United Kingdom
Pre-assignment Details: Total 2968 subjects were enrolled of which 14 subjects were not randomized and were therefore removed from the study (2 subjects withdrew consent and 11 subjects were withdrawn due to inappropriate enrollment and 1 withdrawn due to protocol violation).
Period: Overall Study
Arm/Group | rMenB+OMV | MenACWY | Control
Started | 979 | 988 | 987
Completed | 796 | 844 | 826
Not Completed | 183 | 144 | 161
Not completed — Withdrawal by Subject | 38 | 31 | 28
Not completed — Lost to Follow-up | 124 | 98 | 123
Not completed — Protocol Violation | 5 | 5 | 6
Not completed — Adverse event or death | 11 | 8 | 3
Not completed — Inappropriate enrollment | 2 | 1 | 0
Not completed — Administrative reason | 1 | 0 | 0
Not completed — Unable to classify | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB+OMV | MenACWY | Control | Total
Number analyzed (Participants) | 979 | 988 | 987 | 2954
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (1.6) | 19.9 (1.6) | 19.8 (1.6) | 19.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 516 | 533 | 547 | 1596
  Male | 463 | 455 | 440 | 1358

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Carriage of Virulent Sequence Types (ST) of Neisseria Meningitidis Group B, One Month After Completion of rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of virulent sequence types (ST) of Neisseria meningitidis group B, one month after completion of rMenB+OMV NZ vaccination. The carriage rate of virulent sequence types (ST) of N. meningitidis group B (genogroupable) in subjects, one month after receiving two doses of rMenB+OMV NZ, as compared to the control group, was reported.
  Virulent ST types are defined as Clonal Complex multi locus sequence typing (MLST) or ST type being the same compared to history data (Clonal Complexes MLST or ST types found to be virulent and causing diseases) from the years 2006 to 2010.
Time Frame: 61 days (31 days after receiving the second injection)
Population: Analysis was done on the modified-intention to treat (MITT) dataset (Pharyngeal carriage), i.e subjects who actually received a study vaccination and provided at least one evaluable swab sample at baseline and after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 8 [6 to 10] | 7 [6 to 9]
  Month 2 (N= 916, 928) | 9 [8 to 12] | 8 [6 to 10]
Statistical Analysis 1: Comparison: rMenB+OMV vs Control; Vaccine Group Odds Ratios for carriage of virulent ST strain of N. meningitidis group B in 4CMenB group as compared to the control group at 1 month after receiving the 2nd rMenB+OMV NZ vaccination; Test type: Superiority or Other; p = 0.3828, Regression, Logistic; Odds Ratio (OR) = 1.185, 95% CI 2-sided [0.809 to 1.737]

2. Primary Outcome: Percentages of Subjects With Combined Carriage of N. Meningitidis Serogroups A, C, W and Y, One Month After MenACWY-CRM Vaccination
Description: The percentage of subjects with combined carriage rate of N. meningitidis serogroups A, C, W and Y in subjects, one month after receiving a single dose of MenACWY-CRM conjugate vaccine as compared to the control group is reported.
Time Frame: 31 days after MenACWY-CRM injection
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 981 | 984
Percentages of subjects
  Baseline | 6 [5 to 8] | 5 [4 to 7]
  Month 1 (N=956, 947) | 6 [5 to 8] | 6 [5 to 8]
Statistical Analysis 1: Comparison: MenACWY vs Control; Vaccine Group Odds Ratios for carriage of combined N. meningitidis serogroups A, C, W, Y in the MenACWY-CRM group compared to Control group at 1 month after receiving 1 injection of MenACWY vaccine; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.840, 95% CI 2-sided [0.555 to 1.273]

3. Secondary Outcome: Percentages of Subjects With Carriage of All ST Types of N. Meningitidis B (Genogroupable) at Different Time Points Following rMenB+OMV NZ Vaccination
Description: The percentage of subjects with carriage of all (virulent + non-virulent) ST types of N. meningitidis B (genogroupable) in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 9 [8 to 11] | 9 [7 to 11]
  1 month post 1st vaccination (Day 31) N=931, 947 | 9 [7 to 11] | 9 [7 to 11]
  1 month post 2nd vaccination (Day 61) N=916, 928 | 11 [9 to 13] | 10 [8 to 12]
  3 months post 2nd vaccination (Day 121) N=860, 885 | 10 [8 to 12] | 10 [8 to 12]
  5 months post 2nd vaccination (Day 181) N=832, 864 | 9 [8 to 12] | 10 [8 to 12]
  11 months post 2nd vaccination (Day 361) N=797,827 | 8 [6 to 10] | 10 [8 to 12]

4. Secondary Outcome: Percentages of Subjects With Carriage of Virulent ST Types of N. Meningitidis Group B at Any Time Point After rMenB+OMV NZ Vaccination
Description: Percentage of subjects with carriage of virulent ST types of N. meningitidis group B (genogroupable) in subjects at different time points of the study point after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 8 [6 to 10] | 7 [6 to 9]
  1 month post 1st vaccination (Day 31) N=931,947 | 8 [6 to 10] | 8 [6 to 10]
  1 month post 2nd vaccination (Day 61) N=916, 928 | 9 [8 to 12] | 8 [6 to 10]
  3 months post 2nd vaccination (Day 121) N=860, 885 | 9 [7 to 11] | 9 [8 to 11]
  5 months post 2nd vaccination (Day 181) N=832,864 | 9 [7 to 11] | 9 [7 to 11]
  11 months post 2nd vaccination (Day 361) N=797,827 | 8 [6 to 10] | 9 [7 to 11]

5. Secondary Outcome: Percentages of Subjects With Carriage of Nonvirulent ST Types of N. Meningitidis Group B at Any Time Point After rMenB+OMV NZ Vaccination
Description: Percentage of subjects with carriage of nonvirulent ST types of N. meningitidis group B (genogroupable) in subjects at different time points of the study point after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 1 [1 to 2] | 1 [1 to 2]
  1 month post 1st vaccination (N=931,947) | 1 [0 to 2] | 1 [0 to 2]
  1 month post 2nd vaccination (N=916,928) | 1 [1 to 2] | 2 [1 to 3]
  3 months post 2nd vaccination (N=860,885) | 1 [0 to 2] | 1 [0 to 2]
  5 months post 2nd vaccination (N=832,864) | 1 [0 to 2] | 1 [0 to 2]
  11 months post 2nd vaccination (N=797,827) | 1 [0 to 1] | 1 [0 to 2]

6. Secondary Outcome: Percentages of Subjects With Carriage of All N.Meningitidis Strain at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentage of subjects with carriage of all N.meningitidis strains combined in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 33 [31 to 37] | 31 [28 to 34]
  1 month post 1st vaccination (N=931, 947) | 34 [31 to 37] | 32 [29 to 35]
  1 month post 2nd vaccination (N=916, 928) | 38 [35 to 41] | 36 [33 to 40]
  3 months post 2nd vaccination (N=860, 885) | 35 [32 to 39] | 36 [33 to 39]
  5 months post 2nd vaccination (N=832, 864) | 34 [30 to 37] | 36 [33 to 40]
  11 months post 2nd vaccination (N=797, 827) | 27 [24 to 30] | 30 [27 to 34]

7. Secondary Outcome: Percentages of Subjects With Carriage of N.Meningitidis ABCWY Genogroups at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of N.meningitidis ABCWY genogroups in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 19 [17 to 22] | 17 [15 to 19]
  1 month post 1st vaccination (N=931, 947) | 19 [17 to 22] | 19 [16 to 21]
  1 month post 2nd vaccination (N=916, 928) | 22 [19 to 25] | 22 [19 to 24]
  3 months post 2nd vaccination (N=860, 885) | 20 [17 to 23] | 22 [19 to 25]
  5 months post 2nd vaccination (N=832, 864) | 19 [17 to 22] | 23 [20 to 26]
  11 months post 2nd vaccination (N=797, 827) | 15 [12 to 17] | 18 [15 to 20]

8. Secondary Outcome: Percentages of Subjects With Carriage of N.Meningitidis ACWY Genogroups at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of N.meningitidis ACWY genogroups in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 10 [8 to 12] | 8 [7 to 10]
  1 month post 1st vaccination (N=931, 947) | 11 [9 to 13] | 10 [8 to 12]
  1 month post 2nd vaccination (N=916, 928) | 11 [9 to 13] | 12 [10 to 14]
  3 months post 2nd vaccination (N=860, 885) | 10 [8 to 12] | 12 [10 to 14]
  5 months post 2nd vaccination (N=832, 864) | 10 [8 to 12] | 13 [11 to 15]
  11 months post 2nd vaccination (N=797, 827) | 7 [5 to 8] | 8 [6 to 10]

9. Secondary Outcome: Percentages of Subjects With Carriage of N.Meningitidis Serogroups A,C,W or Y at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of N.meningitidis serogroups A,C,W or Y in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 7 [6 to 9] | 5 [4 to 7]
  1 month post 1st vaccination (N=931, 947) | 7 [5 to 9] | 6 [5 to 8]
  1 month post 2nd vaccination (N=916, 928) | 7 [5 to 9] | 8 [6 to 10]
  3 months post 2nd vaccination (N=860, 885) | 6 [5 to 8] | 8 [6 to 10]
  5 months post 2nd vaccination (N=832, 864) | 6 [5 to 8] | 9 [7 to 11]
  11 months post 2nd vaccination (N=797, 827) | 5 [4 to 7] | 5 [3 to 7]

10. Secondary Outcome: Percentages of Subjects With Carriage of N.Meningitidis Genogroup Y at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of N.meningitidis genogroup Y in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MIIT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 7 [6 to 9] | 7 [5 to 9]
  1 month post 1st vaccination (N=931, 947) | 9 [7 to 11] | 8 [7 to 10]
  1 month post 2nd vaccination (N=916, 928) | 9 [7 to 11] | 10 [9 to 13]
  3 months post 2nd vaccination (N=860, 885) | 8 [6 to 10] | 10 [8 to 12]
  5 months post 2nd vaccination (N=832, 864) | 8 [7 to 10] | 10 [8 to 13]
  11 months post 2nd vaccination (N=797, 827) | 5 [4 to 7] | 6 [5 to 8]

11. Secondary Outcome: Percentages of Subjects With Carriage of N.Meningitidis Serogroup Y at Different Time Points After rMenB+OMV NZ Vaccination
Description: Percentages of subjects with carriage of N.meningitidis serogroup Y in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 974 | 984
Percentages of subjects
  Baseline | 6 [4 to 7] | 5 [3 to 6]
  1 month post 1st vaccination (N=931, 947) | 6 [4 to 8] | 5 [4 to 7]
  1 month post 2nd vaccination (N=916, 928) | 5 [4 to 7] | 7 [6 to 9]
  3 months post 2nd vaccination (N=860, 885) | 5 [4 to 7] | 7 [5 to 9]
  5 months post 2nd vaccination (N=832, 864) | 6 [4 to 8] | 7 [6 to 9]
  11 months post 2nd vaccination (N=797, 827) | 4 [3 to 6] | 4 [3 to 6]

12. Secondary Outcome: Percentages of Subject With Carriage of N. Meningitidis Genogroups ACWY at Different Time Points After MenACWY-CRM Vaccination
Description: Percentages of subject with carriage of N. meningitidis genogroups ACWY in subjects at different time points of the study after administration of a single dose of MenACWY-CRM conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 981 | 984
Percentages of subjects
  Baseline | 9 [7 to 11] | 8 [7 to 10]
  1 month post 1 dose (N=956, 947) | 10 [8 to 12] | 10 [8 to 12]
  2 months post 1 dose (N=929, 928) | 9 [8 to 12] | 12 [10 to 14]
  4 months post 1 dose (N=884, 885) | 10 [8 to 12] | 12 [10 to 14]
  6 months post 1 dose (N=867, 864) | 11 [9 to 13] | 13 [11 to 15]
  12 months post 1 dose (N=845, 827) | 8 [6 to 10] | 8 [6 to 10]

13. Secondary Outcome: Percentages of Subjects With Carriage of N. Meningitidis Serogroups ACWY at Different Time Points After MenACWY-CRM Vaccination
Description: Percentages of subjects with carriage of N. meningitidis serogroups ACWY in subjects at different time points of the study after administration of a single dose of MenACWY-CRM conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 981 | 984
Percentages of subjects
  Baseline (Day 1) | 6 [5 to 8] | 5 [4 to 7]
  1 month post 1 dose (N=956, 947) | 6 [5 to 8] | 6 [5 to 8]
  2 months post 1 dose (N=929, 928) | 5 [4 to 7] | 8 [6 to 10]
  4 months post 1 dose (N=884, 885) | 6 [5 to 8] | 8 [6 to 10]
  6 months post 1 dose (N=867, 864) | 6 [5 to 8] | 9 [7 to 11]
  12 months post 1 dose (N=845, 827) | 4 [3 to 6] | 5 [3 to 7]

14. Secondary Outcome: Percentages of Subjects With Carriage of N. Meningitidis Genogroup Y at Different Time Points After MenACWY-CRM Vaccination
Description: Percentages of subjects with carriage of N. meningitidis genogroup Y in subjects at different time points of the study after administration of a single dose of MenACWY-CRM conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 981 | 984
Percentages of subjects
  Baseline | 7 [5 to 8] | 7 [5 to 9]
  1 month post 1 dose (N=956, 947) | 7 [6 to 9] | 8 [7 to 10]
  2 months post 1 dose (N=929, 928) | 7 [6 to 9] | 10 [9 to 13]
  4 months post 1 dose (N=884, 885) | 8 [6 to 10] | 10 [8 to 12]
  6 months post 1 dose (N=867, 864) | 9 [7 to 11] | 10 [8 to 13]
  12 months post 1 dose (N=845, 827) | 6 [5 to 8] | 6 [5 to 8]

15. Secondary Outcome: Percentages of Subjects With Carriage of N. Meningitidis Serogroup Y at Different Time Points After MenACWY-CRM Vaccination
Description: Percentages of subjects with carriage of N. meningitidis serogroup Y in subjects at different time points of the study after administration of a single dose of MenACWY-CRM conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 981 | 984
Percentages of subjects
  Baseline | 4 [3 to 6] | 5 [3 to 6]
  1 month post 1 dose (N=956, 947) | 5 [4 to 6] | 5 [4 to 7]
  2 months post 1 dose (N=929, 928) | 4 [3 to 5] | 7 [6 to 9]
  4 months post 1 dose (N=884, 885) | 5 [4 to 7] | 7 [5 to 9]
  6 months post 1 dose (N=867, 864) | 5 [4 to 7] | 7 [6 to 9]
  12 months post 1 dose (N=845, 827) | 4 [3 to 5] | 4 [3 to 6]

16. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of All ST Types of N. Meningitidis Genogroup B at Different Time Points Following rMenB+OMV NZ Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of all ST types of N. meningitidis genogroup B in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 748 | 786
Percentages of subjects
  Baseline non-carrier | 90 [87 to 92] | 91 [89 to 93]
  1 month post 1st vaccination (N=671, 715) | 3 [2 to 5] | 4 [2 to 5]
  1 month post 2nd vaccination (N=650, 687) | 3 [2 to 5] | 2 [1 to 3]
  3 months post 2nd vaccination (N=628, 674) | 1 [0 to 2] | 3 [1 to 4]
  5 months post 2nd vaccination (N=623, 656) | 1 [1 to 3] | 2 [1 to 4]
  11 months post 2nd vaccination (N=614, 642) | 3 [2 to 5] | 3 [2 to 5]
  At 3,5,11 months post 2nd vaccination (N=628,674) | 5 [4 to 7] | 7 [6 to 10]

17. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of Virulent ST Types of N. Meningitidis Genogroup B at Different Time Points Following rMenB+OMV NZ Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of virulent ST types of N. meningitidis genogroup B in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 748 | 786
Percentages of subjects
  Baseline non-carrier | 91 [89 to 93] | 92 [90 to 94]
  1 month post 1st vaccination (N=682, 726) | 3 [2 to 5] | 3 [2 to 5]
  1 month post 2nd vaccination (N=659, 699) | 3 [2 to 5] | 2 [1 to 3]
  3 months post 2nd vaccination (N=638, 686) | 1 [0 to 2] | 2 [1 to 4]
  5 months post 2nd vaccination (N=632, 670) | 1 [1 to 3] | 2 [1 to 3]
  11 months post 2nd vaccination (N=623, 656) | 3 [2 to 5] | 2 [1 to 4]
  At 3,5, 11 months post 2nd vaccination (N=638,686) | 5 [4 to 7] | 6 [5 to 9]

18. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of All N. Meningitidis at Different Time Points Following rMenB+OMV NZ Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of all N. meningitidis in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 748 | 786
Percentages of subjects
  Baseline non-carrier | 77 [74 to 80] | 80 [77 to 83]
  1 month post 1st vaccination (N=578, 627) | 17 [14 to 20] | 18 [15 to 21]
  1 month post 2nd vaccination (N=479, 513) | 14 [11 to 18] | 12 [9 to 15]
  3 months post 2nd vaccination (N=410, 452) | 9 [6 to 12] | 13 [10 to 16]
  5 months post 2nd vaccination (N=374, 395) | 8 [5 to 11] | 9 [6 to 12]
  11 months post 2nd vaccination (N=344, 361) | 11 [8 to 15] | 14 [10 to 18]
  At 3,5, 11 months post 2nd vaccination (N=410,452) | 26 [21 to 30] | 31 [27 to 35]

19. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of N. Meningitidis Genogroups ABCWY at Different Time Points Following rMenB+OMV NZ Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of N. meningitidis genogroups ABCWY in subjects at different time points of the study after administration of two doses of rMenB+OMV NZ conjugate vaccine as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 748 | 786
Percentages of subjects
  Baseline non-carrier | 82 [79 to 85] | 84 [82 to 87]
  1 month post 1st vaccination (N=611, 663) | 9 [7 to 12] | 10 [8 to 13]
  1 month post 2nd vaccination (N=553, 592) | 6 [4 to 8] | 7 [5 to 9]
  3 months post 2nd vaccination (N=519, 551) | 4 [3 to 6] | 7 [5 to 9]
  5 months post 2nd vaccination (N=497, 515) | 5 [3 to 7] | 5 [3 to 7]
  11 months post 2nd vaccination (N=472, 491) | 6 [4 to 8] | 6 [4 to 9]
  At 3,5, 11 months post 2nd vaccination (N=519,551) | 14 [11 to 18] | 17 [14 to 20]

20. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of N. Meningitidis Serogroups ACWY at Different Time-points After MenACWY-CRM Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of N.meningitidis serogroups A,C, W or Y at different time-points in the study after MenACWY-CRM vaccination as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 794 | 786
Percentages of subjects
  Baseline non-carrier | 94 [92 to 96] | 95 [93 to 96]
  1 month post 1st vaccination (N=746, 745) | 4 [3 to 6] | 5 [3 to 6]
  1 month post 2nd vaccination (N=712, 709) | 2 [1 to 3] | 4 [3 to 6]
  3 months post 2nd vaccination (N=701, 680) | 2 [1 to 4] | 3 [2 to 5]
  5 months post 2nd vaccination (N=685, 660) | 3 [2 to 4] | 2 [1 to 3]
  11 months post 2nd vaccination (N=666, 650) | 2 [1 to 3] | 1 [1 to 3]
  1,3,5, 11 months post 2nd vaccination (N=712, 709) | 8 [6 to 11] | 10 [8 to 12]

21. Secondary Outcome: Percentages of Subjects With New Acquisition of Pharyngeal Carriage of N. Meningitidis Serogroup Y at Different Time-points After MenACWY-CRM Vaccination
Description: The percentages of subjects with newly acquired pharyngeal carriage of N.meningitidis serogroup Y at different time-points in the study after MenACWY-CRM vaccination as compared to the control group is reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 794 | 786
Percentages of subjects
  Baseline non-carrier | 95 [94 to 97] | 95 [94 to 97]
  1 month post 1st vaccination (N=758, 749) | 4 [2 to 5] | 4 [3 to 6]
  1 month post 2nd vaccination (N=730, 719) | 1 [1 to 2] | 4 [2 to 5]
  3 months post 2nd vaccination (N=719, 693) | 1 [1 to 3] | 2 [1 to 4]
  5 months post 2nd vaccination (N=709, 678) | 2 [1 to 3] | 1 [1 to 3]
  11 months post 2nd vaccination (N=694, 669) | 2 [1 to 3] | 1 [1 to 3]
  1,3,5, 11 months post 2nd vaccination (N=730, 719) | 6 [5 to 8] | 8 [6 to 10]

22. Secondary Outcome: The Duration of Any Carriage of N.Meningitidis Strains After Vaccination With rMenB+OMV
Description: The duration of carriage of any N.meningitidis strains after receiving two doses of rMenB+OMV compared to that in the control group is reported.
Time Frame: Any post vaccination timepoint (the date of first observation of the carriage and the date of the last observation of the carriage)
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of days
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 440 | 470
Number of days
  Genogroup B All STs (N=152, 160) | 127 [92 to 162] | 146 [112 to 180]
  Genogroup B virulent STs (N=142, 142) | 122 [87 to 157] | 147 [113 to 182]
  All N meningitidis | 193 [176 to 210] | 202 [185 to 219]
  Genogroups ABCWY (N=300, 323) | 143 [122 to 164] | 162 [141 to 183]
  Serogroups ACWY (N=131, 142) | 104 [79 to 129] | 113 [87 to 138]
  Serogroup Y (N=106, 123) | 106 [79 to 132] | 117 [91 to 144]

23. Secondary Outcome: The Duration of Carriage of Any N. Meningitidis Strain After Vaccination With MenACWY-CRM
Description: The duration of carriage of any N meningitidis strain after receiving one dose MenACWY-CRM as compared to that in control group is reported.
Time Frame: Any time post vaccination (the date of first observation of the carriage and the date of the last observation of the carriage)
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of days
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 138 | 142
Number of days
  Serogroups ACWY | 88 [62 to 114] | 113 [87 to 138]
  Serogroup Y (N=110, 123) | 86 [59 to 114] | 117 [91 to 144]

24. Secondary Outcome: The Duration of Carriage After New Acquisition N.Meningitidis Strains Following Vaccination With rMenB+OMV Vaccine
Description: The duration of carriage after new acquisition of N.meningitidis strains after receiving two doses of rMenB+OMV vaccine compared to that in the control group is reported.
Time Frame: as for outcome 22
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of days
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 271 | 312
Number of days
  Genogroup B All STs (N=76, 89) | 82 [44 to 120] | 107 [71 to 142]
  Genogroup B virulent STs (N=77, 82) | 80 [42 to 117] | 107 [70 to 143]
  All N meningitidis | 158 [135 to 181] | 165 [142 to 188]
  Genogroups ABCWY (N=165, 201) | 121 [96 to 146] | 146 [122 to 170]
  Serogroups ACWY (N=75, 102) | 111 [79 to 143] | 120 [89 to 151]
  Serogroup Y (N=61, 87) | 111 [76 to 146] | 120 [87 to 153]

25. Secondary Outcome: The Duration of Carriage After New Acquisition N.Meningitidis Strains Following Vaccination With MenACWY Vaccine
Description: The duration of carriage after new acquisition of N.meningitidis strains after receiving one dose of MenACWY-CRM vaccine compared to that in the control group is reported.
Time Frame: as for outcome 22
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of days
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 90 | 102
Number of days
  Serogroups ACWY | 90 [57 to 123] | 120 [89 to 151]
  Serogroup Y (N=74, 87) | 87 [52 to 122] | 120 [87 to 153]

26. Secondary Outcome: Percentages of Subjects With N. Meningitidis Carriage of Virulent ST of Group B, Stratified by Pre-vaccination hSBA Titer After rMenB+OMV NZ Vaccination
Description: The percentages of subjects with N. meningitidis Virulent ST of serogroup B, at different time points of the study, in subjects stratified by pre-vaccination hSBA (<4 and ≥4) titers after administration of two doses of rMenB+OMV NZ vaccine as compared to the control group is reported.
  The serum bactericidal antibodies directed against N.meningitides serogroups, are measured by Serum Bactericidal Assay using human complement (hSBA).
  H44/76, 5/99 and NZ98/254 are strains in serogroup B.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | rMenB+OMV | Control
Number analyzed (Participants) | 133 | 31
Percentage
  Baseline hSBA < 4 (H44/76) (N=60,19) | 0 [0 to 6] | 0 [0 to 18]
  1month post 1st dose; hSBA<4(H44/76) (N=60, 18) | 3 [0 to 12] | 0 [0 to 19]
  1month post 2nd dose; hSBA<4(H44/76) (N=60, 18) | 7 [2 to 16] | 0 [0 to 19]
  3months post 2nd dose; hSBA<4(H44/76) (N=56, 17) | 4 [0 to 12] | 0 [0 to 20]
  5 months post 2nd dose; hSBA <4(H44/76) (N=56, 17) | 7 [2 to 17] | 0 [0 to 20]
  11 months post 2nd dose;hSBA <4(H44/76) (N=56, 16) | 11 [4 to 22] | 0 [0 to 21]
  Baseline hSBA ≥4 (H44/76) | 10 [5 to 16] | 6 [1 to 21]
  1month post 1st dose; hSBA ≥4 (H44/76) (N=130, 30) | 5 [2 to 11] | 10 [2 to 27]
  1 month post 2nd dose;hSBA ≥4 (H44/76) (N=130, 30) | 8 [4 to 14] | 7 [1 to 22]
  3 months post 2nd dose;hSBA ≥4 (H44/76) (N=120,29) | 9 [5 to 16] | 14 [4 to 32]
  5 months post 2nd dose;hSBA ≥4 (H44/76) (N=115,28) | 5 [2 to 11] | 11 [2 to 28]
  11 months post 2nd dose;hSBA ≥4 (H44/76)(N=123,30) | 5 [2 to 10] | 7 [1 to 22]
  Baseline hSBA < 4 (5/99) (N=77, 23) | 5 [1 to 13] | 9 [1 to 28]
  1month post 1st dose; hSBA<4 (5/99) (N=77, 22) | 4 [1 to 11] | 9 [1 to 29]
  1 month post 2nd dose;hSBA <4 (5/99) (N=77, 22) | 6 [2 to 15] | 0 [0 to 15]
  3 months post 2nd dose;hSBA <4 (5/99) (N=71, 21) | 4 [1 to 12] | 10 [1 to 30]
  5 months post 2nd dose;hSBA <4 (5/99) (N=68, 21) | 3 [0 to 10] | 10 [1 to 30]
  11 months post 2nd dose;hSBA <4(5/99) (N=71, 20) | 7 [2 to 16] | 5 [0 to 25]
  Baseline hSBA ≥4 (5/99) (N=116, 27) | 8 [4 to 14] | 0 [0 to 13]
  1month post 1st dose; hSBA ≥4 (5/99) (N=113, 26) | 5 [2 to 11] | 4 [0.097 to 20]
  1 month post 2nd dose;hSBA ≥4 (5/99) (N=113, 26) | 8 [4 to 15] | 8 [1 to 25]
  3 months post 2nd dose;hSBA ≥4 (5/99) (N=105, 25) | 10 [5 to 17] | 8 [1 to 26]
  5 months post 2nd dose;hSBA ≥4 (5/99) (N=103, 24) | 8 [3 to 15] | 4 [0 to 21]
  11 months post 2nd dose;hSBA ≥4(5/99) (N=108, 26) | 6 [3 to 13] | 4 [0.097 to 20]
  Baseline hSBA < 4 (NZ98/254) (N=83, 31) | 2 [0 to 8] | 6 [1 to 21]
  1month post 1st dose; hSBA<4(NZ98/254) (N=81, 30) | 4 [1 to 10] | 7 [1 to 22]
  1month post 2nd dose; hSBA<4 (NZ98/254) (N=81, 30) | 4 [1 to 10] | 0 [0 to 12]
  3 months post 2nd dose;hSBA <4 (NZ98/254)(N=75,29) | 3 [0 to 9] | 3 [0.087 to 18]
  5 months post 2nd dose;hSBA <4 (NZ98/254)(N=70,29) | 3 [0 to 10] | 3 [0.087 to 18]
  11 months post 2nd dose;hSBA <4(NZ98/254)(N=75,28) | 11 [5 to 20] | 4 [0.09 to 18]
  Baseline hSBA ≥4 (NZ98/254) (N=110, 19) | 10 [5 to 17] | 0 [0 to 18]
  1month post 1st dose; hSBA ≥4 (NZ98/254)(N=109,18) | 6 [2 to 12] | 6 [0 to 27]
  1 month post 2nd dose;hSBA ≥4 (NZ98/254)(N=109,18) | 10 [5 to 17] | 11 [1 to 35]
  3 months post 2nd dose;hSBA ≥4(NZ98/254)(N=101,17) | 11 [6 to 19] | 18 [4 to 43]
  5 months post 2nd dose;hSBA ≥4(NZ98/254)(N=101,16) | 8 [3 to 15] | 13 [2 to 38]
  11 months post 2nd dose;hSBA≥4(NZ98/254)(N=104,18) | 4 [1 to 10] | 6 [0 to 27]

27. Secondary Outcome: Percentages of Subjects With N. Meningitidis Carriage of Serogroup Y After MenACWY-CRM Vaccination, Stratified by Pre-vaccination hSBA Titers
Description: The prevalence of carriage of N. meningitidis serogroup Y, at different time points of the study, in subjects stratified by pre-vaccination hSBA (<8 and ≥8) titers, after administration of one dose of MenACWY-CRM vaccine as compared to the control group is reported.
Time Frame: Up to 12 months after vaccination
Population: Analysis was done on the MITT dataset (Pharyngeal carriage)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 152 | 154
Percentages of subjects
  Baseline hSBA <8 (MenY) (N=42, 44) | 0 [0 to 8] | 0 [0 to 8]
  1month post 1st dose; hSBA <8 (MenY) (N=39, 40) | 0 [0 to 9] | 3 [0.063 to 13]
  1 month post 2nd dose;hSBA <8 (MenY) (N=39, 40) | 0 [0 to 9] | 0 [0 to 9]
  3 months post 2nd dose;hSBA <8 (MenY) (N=36, 37) | 0 [0 to 10] | 3 [0.068 to 14]
  5 months post 2nd dose;hSBA <8 (MenY) (N=36, 36) | 0 [0 to 10] | 6 [1 to 19]
  11 months post 2nd dose;hSBA <8 (MenY) (N=34, 35) | 3 [0.074 to 15] | 6 [1 to 19]
  Baseline hSBA ≥8 (MenY) | 6 [3 to 11] | 6 [3 to 11]
  1month post 1st dose; hSBA ≥8 (MenY) (N=146,151) | 6 [3 to 11] | 5 [2 to 10]
  1 month post 2nd dose;hSBA ≥8 (MenY) (N=143, 149) | 5 [2 to 10] | 5 [2 to 10]
  3 months post 2nd dose;hSBA ≥8 (MenY) (N=131, 139) | 8 [4 to 14] | 7 [4 to 13]
  5 months post 2nd dose;hSBA ≥8 (MenY) (N=130, 134) | 9 [5 to 16] | 5 [2 to 10]
  11 months post 2nd dose;hSBA ≥8 (MenY) (N=129,135) | 4 [1 to 9] | 3 [1 to 7]

28. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥1:4 Against N. Meningitidis Serogroup B After rMenB+OMV NZ or MenACWY-CRM Vaccination Compared to Control Group
Description: The percentages of subjects with hSBA titers ≥1:4 against the three strains of N. meningitidis B, after rMenB+OMV NZ or MenACWY-CRM vaccination at different time points of the study as compared to the control group are reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset) i.e all enrolled subjects who actually received a study vaccination, provided at least one evaluable serum sample after vaccination and whose assay result was available for at least one serogroup.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 193 | 49 | 50
Percentages of subjects
  Baseline H44/76 | 69 [62 to 75] | 71 [57 to 83] | 62 [47 to 75]
  1 month post 2nd dose (H44/76) (N=189, 45, 48) | 100 [98 to 100] | 76 [60 to 87] | 63 [47 to 76]
  3 months post 2nd dose (H44/76) (N=173, 40, 46) | 99 [97 to 100] | 73 [56 to 85] | 65 [50 to 79]
  5 months post 2nd dose (H44/76) (N=169, 43, 45) | 100 [98 to 100] | 74 [59 to 86] | 67 [51 to 80]
  11 months post 2nd dose (H44/76) (N=177, 41, 46) | 95 [91 to 98] | 76 [60 to 88] | 70 [54 to 82]
  Baseline 5/99 | 60 [53 to 67] | 45 [31 to 60] | 54 [39 to 68]
  1 month post 2nd dose (5/99) (N=189, 45, 48) | 100 [98 to 100] | 40 [26 to 56] | 58 [43 to 72]
  3 months post 2nd dose (5/99) (N=173, 40, 46) | 99 [97 to 100] | 49 [33 to 65] | 53 [38 to 68]
  5 months post 2nd dose (5/99) (N=169, 43, 45) | 99 [97 to 100] | 49 [33 to 65] | 53 [38 to 68]
  11 months post 2nd dose (5/99) (N=177, 41, 46) | 97 [94 to 99] | 51 [35 to 67] | 63 [48 to 77]
  Baseline NZ98/254 | 57 [50 to 64] | 53 [38 to 67] | 38 [25 to 53]
  1 month post 2nd dose (NZ98/254) (N=189, 45, 48) | 99 [97 to 100] | 53 [38 to 68] | 44 [29 to 59]
  3 months post 2nd dose (NZ98/254) (N=173, 40, 46) | 93 [88 to 96] | 48 [32 to 64] | 48 [33 to 63]
  5 months post 2nd dose (NZ98/254) (N=169, 43, 45) | 91 [85 to 94] | 58 [42 to 73] | 42 [28 to 58]
  11 months post 2nd dose (NZ98/254) (N=177, 41, 46) | 85 [79 to 90] | 66 [49 to 80] | 43 [29 to 59]

29. Secondary Outcome: The hSBA Geometric Mean Titers Against N. Meningitidis Serogroup B, After rMenB+OMV NZ or MenACWY-CRM Vaccination Compared to Control Group.
Description: The hSBA Geometric Mean Titers (GMTs) against the three strains of N. meningitidis serogroup B, after rMenB+OMV NZ or MenACWY-CRM vaccination at different time points of the study as compared to the control group are reported.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 193 | 49 | 50
Titers
  Baseline H44/76 | 11 [8.74 to 14] | 11 [6.59 to 18] | 9.42 [5.73 to 15]
  1 month post 2nd dose (H44/76) (N=189, 45, 48) | 229 [192 to 274] | 11 [7.92 to 16] | 10 [7.18 to 15]
  3 months post 2nd dose (H44/76) (N=173, 40, 46) | 144 [116 to 178] | 9.07 [5.79 to 14] | 11 [7.07 to 16]
  5 months post 2nd dose (H44/76) (N=169, 43, 45) | 111 [89 to 138] | 12 [7.57 to 18] | 12 [7.62 to 18]
  11 months post 2nd dose (H44/76) (N=177, 40, 46) | 68 [54 to 84] | 14 [8.84 to 22] | 14 [8.97 to 21]
  Baseline 5/99 | 6.44 [5.1 to 8.13] | 3.12 [1.97 to 4.95] | 5.49 [3.47 to 8.67]
  1 month post 2nd dose (5/99) (N=189, 45, 48) | 424 [355 to 507] | 2.63 [1.83 to 3.79] | 5.62 [3.95 to 8.01]
  3 months post 2nd dose (5/99) (N=173, 40, 46) | 169 [139 to 207] | 2.95 [1.94 to 4.47] | 5.6 [3.8 to 8.26]
  5 months post 2nd dose (5/99) (N=169, 43, 45) | 105 [87 to 128] | 3.36 [2.27 to 4.97] | 5.32 [3.63 to 7.79]
  11 months post 2nd dose (5/99) (N=177, 41, 46) | 55 [45 to 67] | 3.58 [2.37 to 5.4] | 5.98 [4.05 to 8.82]
  Baseline NZ98/254 | 6.15 [4.82 to 7.84] | 4.32 [2.66 to 7] | 4.16 [2.58 to 6.72]
  1 month post 2nd dose (NZ98/254) (N=188, 45, 48) | 99 [80 to 122] | 4.82 [3.11 to 7.47] | 3.88 [2.54 to 5.93]
  3 months post 2nd dose (NZ98/254) (N=172, 40, 46) | 56 [44 to 73] | 4.93 [2.89 to 8.4] | 4.72 [2.87 to 7.76]
  5 months post 2nd dose (NZ98/254) (N=169, 43, 45) | 50 [38 to 66] | 6.5 [3.73 to 11] | 4.67 [2.72 to 8.03]
  11 months post 2nd dose (NZ98/254) (N=176, 41, 44) | 34 [26 to 45] | 7.77 [4.38 to 14] | 6.93 [3.99 to 12]

30. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥1:8 Against N. Meningitidis Serogroup C and Y, After rMenB+OMV NZ or MenACWY-CRM Vaccination Compared to Control Group.
Description: The percentages of subjects with hSBA titers ≥1:8 against N. meningitidis serogroups C and Y, after rMenB+OMV NZ or MenACWY-CRM vaccination at different time points of the study as compared to the control group are reported.
  As serogroup A and W strains were not detected in substantial proportion of subjects during pharyngeal carriage analysis, these serogroups were not tested.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 193 | 194 | 198
Percentages of subjects
  Baseline Men C (N= 49, 194,50) | 90 [78 to 97] | 87 [81 to 91] | 80 [66 to 90]
  1 month post 2nd dose (Men C) (N=48, 182, 48) | 98 [89 to 100] | 99 [96 to 100] | 88 [75 to 95]
  11 months post 2nd dose (Men C) (N=48, 158, 41) | 94 [83 to 99] | 97 [93 to 99] | 88 [74 to 96]
  Baseline Men Y | 72 [65 to 78] | 78 [72 to 84] | 78 [71 to 83]
  1 month post 2nd dose (Men Y) (N=187, 182, 188) | 81 [74 to 86] | 95 [90 to 97] | 82 [76 to 88]
  3 months post 2nd dose (Men Y) (N=173,164,175) | 79 [72 to 85] | 95 [90 to 97] | 82 [75 to 87]
  5 months post 2nd dose (Men Y) (N=170, 165, 170) | 78 [71 to 84] | 92 [87 to 96] | 84 [77 to 89]
  11 months post 2nd dose (Men Y) (N=177, 158, 165) | 77 [71 to 83] | 91 [86 to 95] | 81 [74 to 87]

31. Secondary Outcome: The hSBA Geometric Mean Titers Against N. Meningitidis Serogroup C and Y, After rMenB+OMV NZ or MenACWY-CRM Vaccination Compared to Control Group.
Description: The hSBA antibody titers against N. meningitidis serogroups C and Y after rMenB+OMV NZ or MenACWY-CRM vaccination at different time points of the study as compared to the control group, are reported as GMTs.
  Serogroups A and W were not analysed.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 193 | 194 | 198
Titers
  Baseline Men C (N=49, 194, 50) | 43 [26 to 70] | 50 [39 to 65] | 32 [20 to 53]
  1 month post 2nd dose (Men C) (N=48, 182, 48) | 83 [55 to 126] | 1302 [1050 to 1615] | 37 [24 to 56]
  11 months post 2nd dose (MenC) (N=48, 158, 41) | 59 [38 to 91] | 438 [343 to 560] | 41 [25 to 66]
  Baseline Men Y | 18 [14 to 22] | 19 [15 to 23] | 19 [15 to 23]
  1 month post 2nd dose (Men Y) (N=187, 182, 188) | 26 [21 to 32] | 83 [67 to 103] | 23 [18 to 28]
  3 months post 2nd dose (Men Y) (N=173, 164, 175) | 24 [19 to 30] | 69 [56 to 86] | 22 [17 to 27]
  5 months post 2nd dose (Men Y (N=170, 165, 170) | 23 [19 to 29] | 63 [51 to 78] | 22 [18 to 28]
  11 months post 2nd dose (Men Y) (N=177, 158, 165) | 21 [17 to 26] | 49 [39 to 61] | 22 [17 to 27]

32. Secondary Outcome: Percentages of Subjects With hSBA Seroresponse Against N. Meningitidis Serogroups C and Y After Vaccination With rMenB+OMV NZ or MenACWY-CRM Compared to Control Group.
Description: The percentages of subjects with hSBA seroresponse against N. meningitidis serogroups C and Y, after rMenB+OMV NZ or MenACWY-CRM vaccination as compared to the control group are reported.
  Seroresponse to N. meningitidis serogroups Cand Y is defined as :(1)for subjects with a pre-vaccination hSBA titer < 1:4 to a post-vaccination hSBA titer ≥ 1:8 or (2) for subjects with a pre-vaccination hSBA titer ≥ 1:4, an increase in hSBA titer of at least four times the pre-vaccination titer.
  Analysis was not done for serogroups A and W.
Time Frame: 61 days
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 187 | 181 | 188
Percentages of subjects
  1 month post 2nd dose from day 1(Men C)N=48,181,48 | 8 [2 to 20] | 81 [75 to 87] | 4 [1 to 14]
  1 month post 2nd dose from day 1(Men Y) | 12 [8 to 17] | 44 [37 to 52] | 7 [4 to 12]

33. Secondary Outcome: The hSBA Geometric Mean Titers Against N. Meningitidis Serogroups C and Y in Subjects (Who Have Received a Prior Dose of MenC Vaccine) After Vaccination With MenACWY-CRM in This Study Compared to Control Group
Description: The hSBA geometric mean titers against the N. meningitidis serogroups C and Y in subjects (who have received a prior dose of MenC vaccine) after MenACWY-CRM vaccination at different time points of the study as compared to the control group are reported.
  Analysis was not done for serogroups A and W.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 46 | 26
Titers
  Baseline (Men C) (N=46, 6) | 91 [51 to 160] | 157 [33 to 756]
  1 month post 2nd vaccination (Men C) (N=45, 6) | 1905 [1305 to 2779] | 154 [55 to 434]
  11 months post 2nd vaccination (Men C) (N=45, 6) | 691 [464 to 1028] | 125 [42 to 371]
  Baseline (Men Y) | 21 [13 to 32] | 23 [13 to 41]
  1 month post 2nd vaccination (Men Y) (N=45, 26) | 89 [55 to 142] | 19 [10 to 36]
  3 months post 2nd vaccination (Men Y) (N=42, 25) | 67 [41 to 110] | 20 [11 to 38]
  5 months post 2nd vaccination (Men Y) (N=45, 26) | 65 [41 to 103] | 20 [11 to 37]
  11 months post 2nd vaccination (Men Y) (N=45, 26) | 48 [31 to 76] | 22 [12 to 39]

34. Secondary Outcome: Percentages of Subjects (Who Have Received a Prior Dose of MenC Vaccine) With hSBA Titers ≥1:8 Against N. Meningitidis Serogroups C and Y After Vaccination With MenACWY-CRM in This Study Compared to Control Group.
Description: The percentages of subjects (who have received a prior dose of MenC vaccine) with hSBA titers ≥1:8 against N. meningitidis serogroups C and Y after receiving MenACWY-CRM vaccination in this study as compared to the control group are reported.
  Analysis was not done for serogroups A and W.
Time Frame: Up to 361 days after vaccination
Population: Analysis was done on the MITT dataset (Immunogenicity subset)
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY | Control
Number analyzed (Participants) | 46 | 26
Percentages of subjects
  Baseline (Men C) (N=46,6) | 93 [82 to 99] | 100 [54 to 100]
  1 month post 2nd vaccination (Men C) (N=45, 6) | 100 [92 to 100] | 100 [54 to 100]
  11 months post 2nd vaccination (Men C) (N=45, 6) | 100 [92 to 100] | 100 [54 to 100]
  Baseline (Men Y) | 80 [66 to 91] | 81 [61 to 93]
  1 month post 2nd vaccination (Men Y) (N=45, 26) | 96 [85 to 99] | 77 [56 to 91]
  3 months post 2nd vaccination (Men Y) (N=42, 25) | 95 [84 to 99] | 80 [59 to 93]
  5 months post 2nd vaccination (Men Y) (N=45, 26) | 96 [85 to 99] | 77 [56 to 91]
  11 months post 2nd vaccination (Men Y) (N=45, 26) | 91 [79 to 98] | 77 [56 to 91]

35. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Vaccination With rMenB+OMV NZ or MenACWY-CRM Compared to Control Group
Description: The safety and tolerability of two doses of rMenB+OMV NZ vaccine (Group rMenB+OMV) and one dose of MenACWY-CRM vaccine (Group MenACWY) was assessed in terms of number of subjects with solicited local and systemic adverse events and other adverse events, following vaccination and compared to that of the control group.
Time Frame: Day 1 through day 7 after any vaccination
Population: Analysis was done on the Immunogenicity Subset, Safety Population i.e. all subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: number of subjects
Arm/Group | rMenB+OMV | MenACWY | Control
Number analyzed (Participants) | 190 | 187 | 191
number of subjects
  Any local | 184 | 158 | 139
  Injection site pain (N=190, 186,191) | 181 | 143 | 117
  Injection site erythema (N=190, 186, 191) | 100 | 71 | 61
  Injection site induration (N=190, 186, 191) | 68 | 41 | 21
  Injection site swelling (N=190, 186, 191) | 68 | 31 | 23
  Any systemic | 169 | 133 | 140
  Arthralgia (N=190, 186, 191) | 38 | 27 | 29
  Nausea (N=190, 186, 191) | 36 | 23 | 24
  Malaise (N=190, 186, 191) | 57 | 41 | 46
  Myalgia (N=190, 186, 191) | 155 | 117 | 112
  Headache (N=190, 186, 191) | 71 | 56 | 75
  Rash (N=190, 186, 191) | 9 | 9 | 12
  Fever (≥38°C) (N= 190, 186,191) | 7 | 5 | 7
  Any Other | 64 | 22 | 25
  Temperature (≥40°C) (N= 190, 186, 191) | 0 | 0 | 0
  Antipyretic preventive med. used (N=190, 186, 191) | 20 | 7 | 3
  Antipyretic treatment med. used (N=190, 186, 191) | 55 | 17 | 22

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected from Day1 to day 7 post vaccination; unsolicited AEs were collected throughout the study period (Day 1-Day 361)
Description: The enrolled and safety set populations differ as 11 subjects (5 in rMenB+OMV, 4 in MeACWY and 2 in Control groups) did not receive the study vaccination and therefore did not have any safety data.
Arm/Group | rMenB+OMV | MenACWY | Control
Serious Adverse Events (participants affected / at risk) | 31/974 | 26/984 | 20/985
Other Adverse Events (participants affected / at risk) | 200/974 | 186/984 | 172/985
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB+OMV (N=974) | MenACWY (N=984) | Control (N=985)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Thyroiditis acute (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0
Edema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 3 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diarrhea infectious (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Genital abscess (Infections and infestations) | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 3 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscloskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Carcinoid tumor pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian germ cell cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
IGA Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Pelvic-ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 1
Ligament operation (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB+OMV (N=974) | MenACWY (N=984) | Control (N=985)
Injection site erythema (General disorders) | 102 | 71 | 61
Injection site induration (General disorders) | 68 | 42 | 21
Injection site pain (General disorders) | 182 | 145 | 117
Injection site swelling (General disorders) | 68 | 32 | 23
Malaise (General disorders) | 58 | 43 | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 155 | 119 | 112
Headache (Nervous system disorders) | 82 | 67 | 85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days